CLINICAL TRIAL: NCT01131533
Title: Intraocular Pharmacokinetics of Erythropoietin After Single Intravitreal Injection in Human
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: hallym unuversity medical center, department of ophthalmology
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010_134
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Pharmacokinetics; Erythropoietin
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erythropoietin (Experimental): patients with chronic macular edema associated with diabetic retinopathy
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — vitrectomy following intravitreal erythropoietin

SUMMARY:
The investigators investigate intraocular concentrations and pharmacokinetics of erythropoietin after a single intravitreal injection in humans.

DETAILED DESCRIPTION:
Intravitreal injections of erythropoietin for off-label use have been shown to be beneficial in eyes with diabetic macular edema.However, the pharmacokinetic profile of erythropoietin after intravitreal injection in humans has not yet been determined clearly. The purpose of this study was to determine the intraocular pharmacokinetics of erythropoietin after a single intravitreal injection in a prospective investigation.

ELIGIBILITY:
Inclusion Criteria:

* diabetic macular edema that failed to respond to or recurred after the previous macular focal laser photocoagulation or intravitreal therapy, or both.
* visual acuity worse than 40/200 snellen bisual acuity

Exclusion Criteria:

* Eyes with vitreomacular traction, active proliferative diabetic retinopathy, intraocular inflammation, uncontrolled intraocular pressure , cataract surgery within the past six months, or a prior history of vitreoretinal surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of erythropoietin in aqueous humor | a few seconds
  erythropoietin injections had been performed in our department following standard procedures. In selected cases,vitrectomy was performed one to two days after erythropoietin injection to treat diabetic macular edema.During surgery, aqueous humor samples were obtained via a corneal paracentesis anterior to the limbus at the beginning of the procedure.

SECONDARY OUTCOMES:
Concentration of erythropoietin in vitreous | few minutes
  erythropoietin injections had been performed in our department following standard procedures. In selected cases,vitrectomy was performed one to two days after erythropoietin injection to treat diabetic macular edema.During surgery, vitreous samples were obtained via vitreous cutter at the beginning of the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Sacred Heart Hoapital, Chuncheon, Kangwondo, South Korea

REFERENCES:
- [Result] Li W, Sinclair SH, Xu GT. Effects of intravitreal erythropoietin therapy for patients with chronic and progressive diabetic macular edema. Ophthalmic Surg Lasers Imaging. 2010 Jan-Feb;41(1):18-25. doi: 10.3928/15428877-20091230-03. PMID 20128565
- [Result] Lagreze WA, Feltgen N, Bach M, Jehle T. Feasibility of intravitreal erythropoietin injections in humans. Br J Ophthalmol. 2009 Dec;93(12):1667-71. doi: 10.1136/bjo.2008.156794. Epub 2009 Aug 18. PMID 19692373
- [Result] Song BJ, Cai H, Tsai JC, Chang S, Forbes M, Del Priore LV. Intravitreal recombinant human erythropoietin: a safety study in rabbits. Curr Eye Res. 2008 Sep;33(9):750-60. doi: 10.1080/02713680802366602. PMID 18798078
- [Result] Zhang J, Wu Y, Jin Y, Ji F, Sinclair SH, Luo Y, Xu G, Lu L, Dai W, Yanoff M, Li W, Xu GT. Intravitreal injection of erythropoietin protects both retinal vascular and neuronal cells in early diabetes. Invest Ophthalmol Vis Sci. 2008 Feb;49(2):732-42. doi: 10.1167/iovs.07-0721. PMID 18235022
- [Derived] Lim JW, Han JR. Aqueous humour levels of vascular endothelial growth factor and erythropoietin in patients with diabetic macular oedema before and after intravitreal erythropoietin injection. Clin Exp Ophthalmol. 2011 Aug;39(6):537-44. doi: 10.1111/j.1442-9071.2011.02510.x. Epub 2011 Mar 24. PMID 21819507